CLINICAL TRIAL: NCT06229821
Title: Safety and Efficacy of Intrapulmonary Percussive Ventilation in Preterm Infants
Acronym: IPV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Augusta University (Other)
Responsible Party: Principal Investigator, Michel Garcia Crespo, Principal Investigator, Augusta University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2067921-2
Record Dates: First submitted 2024-01-16; First posted 2024-01-29 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Respiratory Distress Syndrome in Premature Infant

STUDY DESIGN:
Intervention Model Description: Application of Intrapulmonary Percussive Ventilation (IPV) in preterm neonates, older than 14 days, who require mechanical ventilation. IPV will be administered in increasing intervals, for 15 minutes, starting every 6 hours, and ending every 24 hours; for a total of 7 days.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention group (Other)
  Interventions: Device: Intrapulmonary Percussive Ventilation

INTERVENTIONS:
Device: Intrapulmonary Percussive Ventilation — IPV applied at increasing intervals, starting every 6 hours, and ending at every 24 hours, for a total of 7 days.

SUMMARY:
The purpose of this study is to evaluate the benefits and safety of Intrapulmonary Percussive Ventilation in preterm infants. IPV has been demonstrated to be safe, and improve airway secretions clearance and decreased atelectasis in pediatric patients. We aim to evaluate the effects of IPV in preterm infants.

ELIGIBILITY:
INCLUSION CRITERIA

* Premature infants born before 32 weeks of gestation with birth weight less than 1500 grams.
* Infants requiring positive pressure ventilation by 14 days of life. EXCLUSION CRITERIA
* Infants with known or suspected chromosomal anomalies (Trisomy 13, 18, 21)
* Infants with Congenital Diaphragmatic Hernia
* Presence of air leak syndrome (pneumothorax, pneumomediastinum)
* Previous diagnosis of air leak syndrome.

Min Age: 14 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Mechanical ventilation and supplemental oxygen | From the date of starting treatment protocol to 2 weeks after.
  Need for mechanical ventilation and supplemental oxygen administration

SECONDARY OUTCOMES:
Diagnosis of Bronchopulmonary Dysplasia | At 36 weeks gestational age
  Need for mechanical ventilation and supplemental oxygen administration